CLINICAL TRIAL: NCT01642849
Title: Effect of Diet Composition on Weight Change and Metabolic Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-07996-FB; 1-09-CR-32 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2012-07-03; First posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Obesity; Inflammation
Keywords: high protein diet; high carbohydrate diet; weight loss; oxidative stress; inflammation; cardiovascular risk factors
MeSH Terms: conditions — Obesity; Inflammation; Weight Loss | interventions — Diet, High-Protein; Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- high protein diet (Experimental): 12 subjects will be place on a high protein diet
  Interventions: Dietary Supplement: high protein diet; Dietary Supplement: high carbohydrate diet
- high carbohydrate diet (Experimental): 12 subjects will be put on a high carbohydrate diet for 6 months
  Interventions: Dietary Supplement: high carbohydrate diet

INTERVENTIONS:
Dietary Supplement: high protein diet — 6 months on HP diet
  Arms: high protein diet
Dietary Supplement: high carbohydrate diet — 12 subjects will be placed on a hig carbohydrate diet for 6 months

SUMMARY:
This study will assess the effect of high protein (HP) and high carbohydrate (HC) diets on weight loss and other metabolic parameters.

Rationale: The prevalence of obesity is on the rise in the US. The health hazards of obesity have been well established. The detrimental effects of obesity on cardiovascular, metabolic and psychological parameters as well as the excess cost to the national health budget are astounding. One way of treatment and prevention of obesity has been the use of diet and exercise. In the absence of well-established superiority of one diet over another, different scientifically unproven diets are in common use. A palatable diet providing satiety as well as all essential nutrients may go a long way in treating over-weight individuals. Another factor has been the long-term adherence to such weight loss regimens, which in general have been poor. Protein diets have been known to provide greater satiety and reduced energy intake than carbohydrate diets, but definite long-term studies are sparse. For this study the investigators will recruit and study 24 normal, pre-menopausal obese women (12 on HP diet and 12 on HC diet), and compare their weight loss and changes in metabolic parameters between the two diets.

DETAILED DESCRIPTION:
Population: Recruit and study 24 pre-menopausal women with the following inclusion criteria:

Age range 20 yrs to 50 yrs, BMI > 30 kg/m2 to < 55 kg/m2 Fasting glucose < 110 mg/dl and 120 minute OGTT < 170 mg/dl glucose Design: The study is designed to determine the follow

To compare the effects of high protein (HP) versus high carbohydrate (HC) diet during energy restriction on weight loss, body composition (lean and fat body mass) and bone mineral density in a free living out patient setting.

To assess the effects of HP versus HC diets on metabolic parameters including insulin sensitivity, protein and muscle break down, lipoprotein metabolism and basal metabolic rate.

Procedures: SCREENING VISIT 1:Individuals fulfilling the inclusion and exclusion criteria will be invited for the first screening visit (VS1). A brief study overview will be given along with a brief history and physical examination, height and weight measurements and blood drawn for chemistry profile and and Oral Glucose Tolerance Test (OGTT) to determine normal glucose handling.

SCREENING VISIT 2 (VS2):Individuals fulfilling all the criteria will be contacted and invited for a second screening visit (VS2). Block food frequency questionnaire to assess baseline dietary profile will be given along with a pre-study orientation with the help of a nutritionist.

SCREENING VISIT 3 (VS3): At the final screening visit (VS3) the food diary will be reviewed. Individuals will be randomized into one of the two diet groups using a randomization table. Participants will be asked to participate in the additional studies of euglycemic hyperinsulinemic clamp and indirect calorimetry.

Study participants will either follow a HP or a HC diet for 6 months, where all food is supplied to them. Randomization will be performed using a randomization table. HP diet will be based on 30% Kcals from protein, 40% Kcals from carbohydrate (CHO) and 30% Kcals from fat. In contrast, HC diet will comprise 15% Kcals from protein, 55% Kcals from CHO and 30% Kcals from fat. Subjects will come in weekly for their food pick up and weight checks.

ELIGIBILITY:
Inclusion Criteria:

* Age range 20 yrs to 50 yrs,
* BMI > 30 kg/m2 to < 55 kg/m2
* Fasting glucose < 110 mg/dl and 120 minute OGTT < 170 mg/dl glucose

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Effect of Diet Composition on Weight Change and Metabolic Parameters | 6 months on High Protein or High Carbohydrate diet
  Outcome Measures: The effect of a high protein diet or a high carbohydrate diet provided to subjects for 6 months on metabolic parameters.

SECONDARY OUTCOMES:
Effect of Diet Composition on Weight Change and Metabolic Parameters | 6 months on a high protein or high carbohydrate diet
  The effect of a high protein or high carbohydrate diet supplied to subjects for 6 months on weight loss.

CONTACTS AND LOCATIONS:
Overall Officials: Frankie B. Stentz, M.S., Ph.D., Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Stentz FB, Lawson D, Tucker S, Christman J, Sands C. Decreased cardiovascular risk factors and inflammation with remission of type 2 diabetes in adults with obesity using a high protein diet: Randomized control trial. Obes Pillars. 2022 Dec 1;4:100047. doi: 10.1016/j.obpill.2022.100047. eCollection 2022 Dec. PMID 37990670
- [Derived] Stentz FB, Mikhael A, Kineish O, Christman J, Sands C. High protein diet leads to prediabetes remission and positive changes in incretins and cardiovascular risk factors. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1227-1237. doi: 10.1016/j.numecd.2020.11.027. Epub 2020 Dec 8. PMID 33549435